CLINICAL TRIAL: NCT01997931
Title: The Impact of Bispectral Index Monitoring on Sedation Administration in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111/04
Record Dates: First submitted 2005-09-09; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Intensive Care; Mechanically Ventilated Patients; Sedated Patients
Keywords: bispectral index; sedation; intensive care; mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bispectral Index Sedation monitor

SUMMARY:
This prospective randomised controlled trial was designed to assess the effectiveness of the Bispectral Index Sedation (BIS) monitor in supporting clinical, sedation management decisions in mechanically ventilated ICU patients.

The primary hypothesis for the study is that patients with Bispectral Index Sedation (BIS) monitoring will receive less sedation then those receiving standard sedation management.

The secondary hypotheses are:

1. Patients with BIS have fewer ventilation days than those receiving standard sedation management.
2. Level of sedation administered will differ according to the critical care experience and qualification of the nurse.

DETAILED DESCRIPTION:
Patients in intensive care units (ICUs) frequently require sedatives and analgesics as part of therapy. Assessing the appropriate dose of sedative and analgesic drugs can be difficult due to the severity of the patient's illness, inability of the patient to communicate, multiple procedures and transports for investigations and the subjectivity of clinical sedation assessment tools. Poorly assessed and managed levels of sedation can result in over sedation, extended ventilation time and a potentially extended ICU stay.

The BIS monitor is derived from the electroencephalogram and provides a numeric value that represents a measure of cerebral activity. Such an objective measure of the patient's level of sedation may provide a useful tool that will enable nurses to titrate sedation more accurately in an attempt to provide the optimal level of sedation for all ICU patients.

The study will be conducted in the Intensive Care Unit at the Alfred Hospital. This study is designed as a prospective randomised control trial with parallel design. This means that participants' will be randomly allocated into either one of two groups - an intervention or control group. Participant's randomised to the intervention group will receive BIS monitoring. The control group will receive standard ICU sedation assessment and management.

To determine if BIS monitoring is useful in ICU, information will be collected by auditing patient charts and determining the average amounts of sedation medication for each nursing shift. In addition, the years of critical care experience and critical care qualification will be recorded for each nurse managing patients recruited to the study.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and ventilated for at least 24 hours
* Sedated on morphine and midazelam infusions

Exclusion Criteria:

* Intracranial injury
* Status epilepticus
* Facial Burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-09; Primary Completion 2005-06 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Optimised sedation management for patients through the use of BIS monitoring.

SECONDARY OUTCOMES:
Reduction in mechanical ventilation time.
Reduced length of stay in the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy A Weatherburn, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia